CLINICAL TRIAL: NCT07024784
Title: A Phase 1b Dose Escalation and Expansion Study of IMGN151 as Monotherapy and in Combination With Other Anti-Cancer Therapies in Subjects With Gynecologic Cancers
Brief Title: A Study to Assess Change in Disease Activity and Adverse Events in Adult Participants With Gynecologic Cancers Receiving Intravenous Infusion of IMGN151 as Monotherapy or in Combination With Other Therapies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M25-219; 2023-506842-22-00 (Other: EU CT); GOG-3124 (Other: GOG)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Gynecologic Cancers; Platinum-Sensitive Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer (PSOC)
Keywords: Gynecologic Cancers; Platinum-Sensitive Ovarian Cancer; Platinum-Resistant Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer (PSOC); Cancer; IMGN151
MeSH Terms: conditions — Fallopian Tube Neoplasms; Neoplasms | interventions — Carboplatin; Bevacizumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm A: IMGN151 + Carboplatin (For PSOC) (Experimental): Participants will receive IMGN151 in combination with Carboplatin on Day 1 of a 21-day cycle.
  Interventions: Drug: IMGN151; Drug: Carboplatin
- Arm B: IMGN151 + Olaparib (For PSOC) (Experimental): Participants will receive IMGN151 in combination with Olaparib twice a day (BID) on Day 1 of a 21-day cycle.
  Interventions: Drug: IMGN151; Drug: Olaparib
- Arm C: IMGN151 + Bevacizumab (For PSOC or PROC) (Experimental): Participants will receive IMGN151 in combination with Bevacizumab Day 1 of a 21-day cycle.
  Interventions: Drug: IMGN151; Drug: Bevacizumab
- Arm D: IMGN151 Monotherapy (For PSOC) (Experimental): Participants will receive IMGN151 Day 1 of a 21-day cycle.
  Interventions: Drug: IMGN151
- Arm E: IMGN151 Monotherapy (For PROC in China) (Experimental): Participants will receive IMGN151 Day 1 of a 21-day cycle.
  Interventions: Drug: IMGN151
- Arm F: IMGN151 Monotherapy (For PROC in Japan) (Experimental): Participants will receive IMGN151 Day 1 of a 21-day cycle.
  Interventions: Drug: IMGN151

INTERVENTIONS:
Drug: IMGN151 — Intravenous (IV) infusion
Drug: Carboplatin — Intravenous (IV) infusion
  Arms: Arm A: IMGN151 + Carboplatin (For PSOC)
Drug: Bevacizumab — Intravenous (IV) infusion
  Arms: Arm C: IMGN151 + Bevacizumab (For PSOC or PROC)
Drug: Olaparib — Oral Tablet
  Arms: Arm B: IMGN151 + Olaparib (For PSOC)

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess safety and tolerability of IMGN151 when given as monotherapy and in combination with other anti-cancer therapies in adult participants with gynecologic cancers.

IMGN151 is an investigational drug being developed for the treatment of gynecologic cancers. Participants are placed in 1 of 4 groups, called treatment arms. Each group receives a different treatment. Around 377 participants with gynecologic cancers will be enrolled in the study at approximately 50 sites worldwide.

Participants will receive intravenous infusions of IMGN151 as monotherapy or in combination with anti-cancer therapies according to their assigned study arm. In Arm A, participants will receive IMGN151 in combination with carboplatin on Day 1 of each cycle. In Arm B, participants will receive IMGN151 in combination with olaparib, twice a day (BID) on Day 1 of each cycle. In Arm C, participants will receive IMGN151 in combination with bevacizumab on Day 1 of each cycle. In Arm D, participants will receive IMGN151 as monotherapy on Day 1 of each cycle. In Arm E, participants will receive IMGN151 as monotherapy on Day 1 of each cycle. In Arm F, participants will receive IMGN151 as monotherapy on Day 1 of each cycle. The total study duration will be approximately 3 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 or 1
* Participants (except for platinum-sensitive ovarian, fallopian tube, and primary peritoneal cancer (PSOC) participants without disease progression after platinum combination standard of care therapy in Arms B and D) will have ≥ 1 lesion that meets the definition of measurable disease by RECIST v1.1 (radiographically measured by the investigator).
* Participants will have high-grade serous epithelial ovarian, fallopian tube, and primary peritoneal cancers (EOC).
* Participant has completed prior therapy within the specified times below:

  * Systemic antineoplastic therapy within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose of IMGN151.
  * Focal radiation completed ≥ 2 weeks prior to the first dose of study treatment.

Exclusion Criteria:

* Participants with ovarian cancer with histologies including: endometrioid, clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of the above histologies, as well a low-grade or borderline ovarian tumor.
* History of clinically significant medical conditions or any other reason that the investigator determines would interfere with the participant's participation in this study or would make the participant an unsuitable candidate to receive study treatment.
* Prior treatment with FRα-targeting therapy.
* Prior wide-field radiotherapy affecting more than 20% of the bone marrow.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicities (DLTs) | Up to approximately 3 years
  Dose limiting toxicities (DLTs) of IMGN151 when given as monotherapy and in combination with other anti-cancer therapies DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.
Percentage of Participants with Adverse Events (AE) | Up to approximately 3 years
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

SECONDARY OUTCOMES:
Objective Response (OR) | Up to approximately 3 years
  Defined as achieving confirmed response (complete response [CR] + partial response [PR]) assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.
Duration of response (DOR) | Up to approximately 3 years
  Defined as the time from initial response of CR or PR until investigator assessed radiographical PD per RECIST v1.1 or death of any cause, whichever occurs first.
Progression-free survival (PFS) | Up to approximately 3 years
  Defined as the time from the first dose of study treatment until investigator-assessed radiographical PD per RECIST v1.1 or death of any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (7):
- Israel (4):
  - The Chaim Sheba Medical Center /ID# 275997, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 275852, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 276004, Haifa
  - Shaare Zedek Medical Center /ID# 275854, Jerusalem
- Japan (3):
  - Hyogo Cancer Center /ID# 276940, Akashi-shi, Hyōgo
  - National Cancer Center Hospital /ID# 276715, Chuo-Ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 276711, Koto-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-219